CLINICAL TRIAL: NCT04610073
Title: Comparison of the Effect of Interactive Multimedia Versus Illustrated Booklet on Behavior to Prevent Lower Back Pain in Working Nurses in the Hospitals Affiliated to Shiraz University of Medical Sciences.
Brief Title: The Effect of Interactive Multimedia Versus Illustrated Booklet on Behavior to Prevent Lower Back Pain in Working Nurses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nahid Zarifsanaiey (Other)
Responsible Party: Sponsor-Investigator, Nahid Zarifsanaiey, Associate Professor, Shiraz University of Medical Sciences
Organization: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IR.SUMS.REC.1397.1093
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interactive multimedia training (Experimental): the intervention group 1 completed the pretest knowledge, attitude, and behavior questionnaire. Then, interactive multimedia was made available to this group. The questionnaire was completed again by the group, one week after completion of training, and then one month afterward.
  Interventions: Behavioral: Interactive multimedia training and illustrated booklet
- illustrated booklet (Experimental): First, the intervention group 2 completed the pretest knowledge, attitude, and behavior questionnaire. Then, illustrated booklet was made available to this group. The questionnaire was completed again by the group one week after completion of training, and then one month afterward.
  Interventions: Behavioral: Interactive multimedia training and illustrated booklet
- No Intervention (Experimental): In the control group, no intervention was performed. Only before the intervention, one week and one month after the intervention, they completed the knowledge, attitude and behavior questionnaires.
  Interventions: Behavioral: Interactive multimedia training and illustrated booklet

INTERVENTIONS:
Behavioral: Interactive multimedia training and illustrated booklet — The experimental groups conducted interactive multimedia training and illustrated booklet

SUMMARY:
The present study was conducted to compare the effect of interactive multimedia and illustrated booklet methods on knowledge, attitude and improvement of behavior in preventing lower back pain amongst lower back pain amongst nurses.

DETAILED DESCRIPTION:
In this single blind randomized controlled trial, 153 eligible nurses working in hospitals during 2019 were enrolled. The participants were randomly allocated into three parallel groups: interactive multimedia (n=55), illustrated booklet (n= 55), and the control (n= 43). The study samples were blinded to intervention and control groups. A researcher-made questionnaire was completed by the eligible subjects before, after, and four weeks after the intervention to assess their knowledge, attitude and behavior in preventing chronic lower back pain amongst working nurses.

ELIGIBILITY:
Inclusion Criteria:

* Minimum education level of bachelor's degree in nursing
* Employment in governmental hospitals
* Willing to participate in the study and complete the informed consent
* Minimum knowledge of working with computers

Exclusion Criteria:

* Congenital anomalies
* low back pain
* History of back surgery
* History of trauma to the back
* Pregnancy
* Severe osteoporosis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2019-07-28 (Actual); Study Completion 2019-12-29 (Actual)

PRIMARY OUTCOMES:
Behavior of the employed nurses in order to prevent low back pain | 5 weeks
  Researcher made questionnaire for measuring behavior with 19 questions based on a six-point Likert scale.

SECONDARY OUTCOMES:
Knowledge of the employed nurses in order to prevent low back pain | 5 weeks
  A Researcher made questionnaire for measuring knowledge with 10 four-option questions.
Attitude of the employed nurses in order to prevent low back pain | 5 weeks
  A researcher made questionnaire for measuring attitude with 18 questions based on a six-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nahid zarifsanaiey, PhD, Principal Investigator — associate Professor, Virtual school, Shiraz University of Medical Sciences, Shiraz, Iran.
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: Undecided